CLINICAL TRIAL: NCT02462486
Title: Safety and Efficacy of Abicipar Pegol (AGN-150998) in Patients With Neovascular Age-related Macular Degeneration (SEQUOIA Study)
Brief Title: Safety and Efficacy of Abicipar Pegol in Participants With Neovascular Age-related Macular Degeneration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 150998-006; 2014-004580-20 (EudraCT Number); SEQUOIA (Other: Allergan)
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Results first posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — abicipar pegol; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Abicipar Pegol 2 mg (2Q8) (Experimental): Abicipar pegol 2 mg was administered to the study eye by intravitreal injection on Day 1, Week 4, and Week 8, followed by injections every 8 weeks through Week 96. Scheduled visits occurred every 4 weeks. To maintain masking, sham was administered to the study eye at scheduled visits where abicipar was not administered.
  Interventions: Drug: Abicipar Pegol; Other: Sham Procedure
- Abicipar Pegol 2 mg (2Q12) (Experimental): Abicipar pegol 2 mg was administered to the study eye by intravitreal injection on Day 1, Week 4, and Week 12, followed by injections every 12 weeks through Week 96. Scheduled visits occurred every 4 weeks. To maintain masking, sham was administered to the study eye at scheduled visits where abicipar was not administered.
  Interventions: Drug: Abicipar Pegol; Other: Sham Procedure
- Ranibizumab (rQ4) (Active Comparator): Ranibizumab (Lucentis®) was administered to the study eye by intravitreal injection every 4 weeks from Day 1 through Week 96.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Abicipar Pegol — Abicipar pegol intravitreal injection.
  Other Names: AGN-150998
  Arms: Abicipar Pegol 2 mg (2Q12); Abicipar Pegol 2 mg (2Q8)
Drug: Ranibizumab — Ranibizumab intravitreal injection.
  Other Names: Lucentis®
  Arms: Ranibizumab (rQ4)
Other: Sham Procedure — Sham injection.
  Arms: Abicipar Pegol 2 mg (2Q12); Abicipar Pegol 2 mg (2Q8)

SUMMARY:
This is a safety and efficacy study of abicipar pegol in participants with neovascular age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of age-related macular degeneration in at least 1 eye
* Best corrected visual acuity of 20/40 to 20/320 in the study eye
* Best corrected visual acuity of 20/200 or better in the non-study eye

Exclusion Criteria:

* History of vitrectomy, macular surgery, or glaucoma surgery in the study eye
* Cataract or refractive surgery in the study eye within the last 3 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 949 (Actual)
Dates: Start 2015-06-25 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2019-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Li, Study Director — Allergan
Locations (187):
- United States (73):
  - Eye Foundation Hospital, Birmingham, Alabama
  - Retinal Consultants of Arizona, Gilbert, Arizona
  - Barnet Dulaney Perkins Eye Center - Phoenix, Phoenix, Arizona
  - Retina Centers, PC, Tucson, Arizona
  - Northwest Arkansas Retina Associates, Springdale, Arkansas
  - Win Retina, Arcadia, California
  - Retina Institute of California, Arcadia, California
  - Retinal Diagnostic Center, Campbell, California
  - Specialty Eye Care Medical Center, Inc., Glendale, California
  - University of California at Irvine Gavin Herbert Eye Institute, Irvine, California
  - Retina Associates of Orange County, Laguna Hills, California
  - South Coast Retina Center, Long Beach, California
  - East Bay Retina Consultants, Inc., Oakland, California
  - San Diego Retina Associates, Oceanside, California
  - Southern California Desert Retina Consultants, Palm Desert, California
  - California Eye Specialist Medical Group, Pasadena, California
  - Retina Consultants, San Diego, Poway, California
  - Retina Consultants of Southern California, Redlands, California
  - Kaiser Permanente Riverside Medical Center, Riverside, California
  - UC Davis Medical Center, Department of Ophthalmology, Sacramento, California
  - Retinal Consultants Medical Group, Inc., Sacramento, California
  - West Coast Retina Medical Group, San Francisco, California
  - Pacific Eye Associates, San Francisco, California
  - The Eye Associates, Bradenton, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Retina Macula Specialists of Miami, Miami, Florida
  - MedEye Associates, Miami, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Retina Associate of Florida, P.A., Tampa, Florida
  - Retina Vitreous Associates of Florida, Tampa, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - DuPage Medical Group, Downers Grove, Illinois
  - Kovach Eye Institute, Elmhurst, Illinois
  - University Retina and Macula Associates, Oak Forest, Illinois
  - Wheaton Eye Clinic, Clinical Research Center, LLC, Wheaton, Illinois
  - Sabates Eye Centers, Leawood, Kansas
  - Paducah Retinal Center, Paducah, Kentucky
  - The Retina Care Center, Baltimore, Maryland
  - Cumberland Valley Retina Consultants, P.C., Hagerstown, Maryland
  - Vitreo-Retinal Associates, Pc, Worcester, Massachusetts
  - Retina Specialists of Michigan, Grand Rapids, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Retina Center of New Jersey, LLC, Bloomfield, New Jersey
  - Delaware Valley Retina Associates, Lawrenceville, New Jersey
  - Long Island Vitreoretinal Consultants, Hauppauge, New York
  - Maculacare - New York, New York, New York
  - Retina Vitreous Surgeons of Central NY, PC, Syracuse, New York
  - Western Carolina Retinal Associates, PA, Asheville, North Carolina
  - Charlotte Eye Ear Nose & Throat Associates, PA, Charlotte, North Carolina
  - Retina Associates of Cleveland, Inc, Beachwood, Ohio
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Midwest Retina, Inc., Dublin, Ohio
  - Retina & Vitreous Center SO, PC, Ashland, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - Pennsylvania Retina Specialists, P.C., Camp Hill, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Austin Retina Associates, Austin, Texas
  - Retina and Vitreous of Texas, Beaumont, Texas
  - The University of Texas Medical Branch, Galveston, Texas
  - Premiere Retina Specialists, Midland, Texas
  - Retina Associates of South Texas, PA, San Antonio, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - University of Utah, John Moran Eye Center, Salt Lake City, Utah
  - Virginia Eye Consultants, Norfolk, Virginia
  - Wagner Macula and Retina Center, Virginia Beach, Virginia
  - Vitreoretinal Associates of Washington, Bellevue, Washington
  - Spokane Eye Clinical Research, Spokane, Washington
  - West Virginia University Eye Institute, Morgantown, West Virginia
- Australia (6):
  - Save Sight Institute, University of Sydney Eye Hospital, Sydney, New South Wales
  - Sydney Retina Clinic and Day Surgery, Sydney, New South Wales
  - Sydney West Retina, Westmead, New South Wales
  - Centre for Eye Research Australia, East Melbourne, Victoria
  - Specialist Eye Group, Glen Waverley, Victoria
  - Lions Eye Institute, Nedlands, Western Australia
- Brazil (5):
  - Centro Brasileiro de Cirurgia de Olhos - CBCO, Goiânia, Goiás
  - Instistuto da Visao - Hospital de Olhos Ltda, Belo Horizonte, Minas Gerais
  - Hospital Oftalmologico de Sorocaba, Sorocaba, São Paulo
  - Clinica de Olhos Dr. Suel Abujamra, São Paulo
  - Instituto Da Visao UNIFESP EPM (Universidade Federal de Sao Paulo - Escola Paulista de Medicina), São Paulo
- Canada (5):
  - Calgary Retina Consultants, Calgary, Alberta
  - St Joseph's Health Care London - Ivey Eye Institute, London, Ontario
  - Canadian Centre for Advanced Eye Therapeutics Inc, Mississauga, Ontario
  - University of Ottawa Eye Institute, Ottawa, Ontario
  - Toronto Retina Institute, Toronto, Ontario
- Denmark (2):
  - Rigshospitalet-Glostrup, Glostrup Municipality, Capital Region
  - Odense University Hospital, Odense, Region Syddanmark
- Hungary (9):
  - Magyar Honvedseg Egeszegugyi Kozpont, Budapest
  - Semmelweis University, Budapest
  - Bajcsy-Zsilinszky Hospital, Budapest
  - Szent Imre Teaching Hospital, Budapest
  - Budapest Retina Associates Kft., Budapest
  - University of Debrecen, Medical Center, Debrecen
  - Ganglion Medical Centre, Pécs
  - University of Szeged, Szeged
  - Markusovszki Teaching Hospital, Szombathely
- Italy (13):
  - Ospedale Clinicizzato, Chieti, Abruzzo
  - Clinica Oculistica, Ospedale Santa Maria della Misericordia, Udine, Friuli Venezia Giulia
  - Eye Clinic - Fondazione IRCCS, Milan, Lombardy
  - Clinica Oculistica- Dipartimento di Scienze Cliniche Universita di Milano, Milan, Lombardy
  - Ospedale Molinette, Turin, Piedmont
  - Azienda Ospedaliero-Universitaria Careggi - SOD Oculistica, Dipartimento di Chirurgia e Medicina Traslazionale, Florence, Tuscany
  - Azienda Universitaria Ospedaliera Pisana, Ospedale "Nuovo S.Chiara" Cisanello, Pisa, Tuscany
  - IRCCS - Istuto di Recovero e Cura a Carattere Scientifico, Verona, Vento
  - A.O.U. Policlinico Sant Orsola Malpighi Pad1, 4Piano, Studio Medici via Pelagio Palagi 9, Bologna
  - Clinica Oculistica DINOGMI Universita di Genova, Genova
  - IRCCS Ospedale San Raffaele, Milan
  - Policlinico Agostino Gemelli, Roma
  - Fondazione G.B. Bietti-IRCCS, Roma
- Japan (32):
  - Aichi Medical University Hospital, Nagakute, Aichi-ken
  - Japan Community Health Care Organization Chukyo Hospital, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Kameda Clinic, Kamogawa, Chiba
  - Toho University Sakura Medical Center, Sakura, Chiba
  - Juntendo University Urayasu Hospital, Urayasu, Chiba
  - Ogaki Tokushukai Hospital, Ōgaki, Gifu
  - Kimura Eye And Internal Medicine Hospital, Kure, Hiroshima
  - Sapporo City General Hospital, Sapporo, Hokkaido
  - Hyogo Prefectural Amagasaki Hospital General Medical Center, Amagasaki, Hyōgo
  - Tokyo Medical University Ibaraki Medical Center, Inashiki, Ibaraki
  - Mito Kyodo General Hospital, Mito, Ibaraki
  - Otakeganka Tsukimino Clinic, Yamato, Kanagawa
  - Kikuna Yuda Eye Clinic, Kanagawa, Kanto
  - Mie University Hospital, Tsu, Mie-ken
  - Iida Municipal Hospital, Iida, Nagano
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Nihon University Hospital, Chiyoda City, Tokyo
  - Chofu Eye Clinic, Chōfu, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Hachiōji, Tokyo
  - Takeuchi Eye Clinic, Taitō City, Tokyo
  - Kyushu University Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Kokura Kinen Hospital, Kitakyushu
  - Ideta Eye Hospital, Kumamoto
  - The Japanese Red Cross Nagasaki Genbaku Hospital, Nagasaki
  - Nara Medical University Hospital, Nara
  - Medical Corporation Jinshikai Nishi Eye Hospital, Osaka
  - Musashi Dream Clinic, Osaka
  - Tane Memorial Eye Hospital, Osaka
  - Tokyo Women's Medical University Hospital, Tokyo
- Netherlands (4):
  - Elisabeth Hospital, Tilburg, North Brabant
  - Academic Medical Center, Amsterdam, North Holland
  - Oogziekenhuis Rotterdam, Rotterdam, North Holland
  - Leiden University Medical Center, Leiden, South Holland
- Macula D&T Eye Center, San Isidro, Lima region, Peru
- Poland (5):
  - Optimum Profesorskie Centrum Okulistyki, Gdansk
  - Klinika Okulistyczna Jasne Blonia, Lodz
  - Centrum Diagnostyki i Mikrochirurgii, Olsztyn
  - Retina Eye Hospital, Warsaw
  - Uniwersytecki Szpital Kliniczny, Wroclaw
- Russia (2):
  - Scientific Research Institute of Ocular Diseases of RAMS, Moscow
  - S. Fyodorov Eye Microsurgery Federal State Institution, Moscow
- South Africa (3):
  - Pasteur Medical Centre, Bloemfontein
  - Dr Actons Privat Practice, Cape Town
  - Pretoria Eye Institute, Private Practice, Pretoria
- Taiwan (5):
  - Department of Ophthalmology Kaohsiung Veterans General Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Department of Ophthalmology National Taiwan University Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Chang Gung Medical Foundation, Linkou Branch, Taoyuan District
- Turkey (Türkiye) (2):
  - Ankara Uni Med Fac, Ankara
  - Dokuz Eylul Uni Med Fac, Izmir
- United Kingdom (20):
  - Frimley Park Hospital, Frimley, Camberley
  - Royal Derby Hospital, Derby, Derbyshire
  - ESNEFT Essex County Hospital, Colchester, Essex
  - University Hospital Southampton, Southampton, Hampshire
  - Oxford Eye Hospital, John Radcliffe Hospital, Oxford, Headington
  - Royal Liverpool University Hospital, Liverpool, North West England
  - Royal Surrey Hospital, Guildford, South East
  - Heart of England NHS Foundation Trust, Good Hope Hospital, Sutton Coldfield, Staffordshire
  - University Hospital of Wales, Cardiff, Wales
  - Bradford Royal Infirmary (BRI), Bradford, West Yorkshire
  - Sheffield Teaching Hospitals, Sheffield, Yorkshire
  - Barnet Hospital, Barnet
  - Bristol Eye Hospital, Bristol
  - University Hospital Aintree, Liverpool
  - Moorfields Eye Hospital, London
  - Barnet Royal Free Hospital, London
  - King's College Hospital, London
  - Royal Victoria Infirmary, Newcastle
  - Hospital of St. Cross, Rugby
  - City Hospitals Sunderland NHS, Sunderland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abicipar Pegol 2 mg (2Q8) | Abicipar Pegol 2 mg (2Q12) | Ranibizumab (rQ4)
Started | 316 | 315 | 318
Completed | 222 | 223 | 266
Not Completed | 94 | 92 | 52
Not completed — Screen Failure:Missed Exclusion Criteria | 1 | 1 | 3
Not completed — Adverse Event | 53 | 48 | 21
Not completed — Lack of Efficacy | 6 | 12 | 3
Not completed — Lost to Follow-up | 3 | 4 | 2
Not completed — Withdrawal by Subject | 25 | 22 | 19
Not completed — Protocol Violation | 3 | 1 | 1
Not completed — Reason not Specified | 3 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Abicipar Pegol 2 mg (2Q8) | Abicipar Pegol 2 mg (2Q12) | Ranibizumab (rQ4) | Total
Number analyzed (Participants) | 316 | 315 | 318 | 949
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.9 (8.6) | 76.2 (8.3) | 75.9 (8.4) | 76.0 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179 | 174 | 185 | 538
  Male | 137 | 141 | 133 | 411
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 266 | 266 | 264 | 796
  Black | 2 | 4 | 3 | 9
  Asian | 39 | 35 | 41 | 115
  Hispanic | 7 | 8 | 9 | 24
  Other | 2 | 0 | 0 | 2
  Not Reported | 0 | 1 | 1 | 2
  Unknown | 0 | 1 | 0 | 1
Best Corrected Visual Acuity (BCVA) for Per Protocol Population [Mean (Standard Deviation); unit: letters] — BCVA was measured using an eye chart and is reported as number of letters read correctly using Early Treatment of Diabetic Retinopathy Study (ETDRS) Scale (0 to 100 letters) in study eye. Lower number of letters read correctly, worse the vision. Study eye: eye that meets entry criteria. If both eyes met all of entry criteria, eye with worse BCVA at baseline (Day 1) was selected. If values for both eyes were identical, participant selected non-dominant eye, or else right eye was selected. Population: Per Protocol (PP) population included all randomized and treated participants without any protocol deviations that impacted the primary efficacy variable and with treatment compliance to represent the intended regimen adequately.
  letters
    number analyzed (Participants) | 267 | 265 | 299 | 831
    (all) | 57.8 (12.1) | 56.3 (12.5) | 57.0 (12.3) | 57.0 (12.3)
BCVA for ITT Population [Mean (Standard Deviation); unit: letters] — BCVA was measured using an eye chart and is reported as number of letters read correctly using Early Treatment of Diabetic Retinopathy Study (ETDRS) Scale (0 to 100 letters) in study eye. Lower number of letters read correctly, worse the vision. Study eye: eye that meets entry criteria. If both eyes met all of entry criteria, eye with worse BCVA at baseline (Day 1) was selected. If values for both eyes were identical, participant selected non-dominant eye, or else right eye was selected.
  letters | 57.2 (12.3) | 56.4 (12.5) | 57.1 (12.3) | 56.9 (12.4)
Central Retinal Thickness (CRT) [Mean (Standard Deviation); unit: microns] — CRT was assessed using spectral domain optical coherence tomography (SD-OCT), a non-invasive diagnostic system that provides high-resolution imaging sections of retina. SD-OCT was performed in study eye after pupil dilation.Study eye was defined as the eye that meets the entry criteria. If both the eyes met all of the entry criteria, the eye with worse BCVA at baseline (Day 1) was selected. If BCVA values for both eyes were identical then participant had to select the non-dominant eye, or else right eye was selected as study eye. Population: Number analyzed is the number of participants with data available at the Baseline.
  microns
    number analyzed (Participants) | 316 | 314 | 318 | 948
    (all) | 380.3 (117.9) | 378.2 (123.8) | 382.4 (130.3) | 380.3 (124.0)
National Eye Institute Visual Functioning Questionnaire-25 (NEI-VFQ-25) [Mean (Full Range); unit: score on a scale] — NEI-VFQ-25 consists of 25 vision-targeted questions that represent 11 vision-related quality of life subscales and one general health item. Responses of individual participants were recorded as scores that ranged between 0 (worst) to 100 (best vision related function) with higher scale indicating better vision related function. The overall composite score is then calculated by averaging over all 11 vision-targeted subscale scores, excluding the general health score. Overall composite score was calculated based on mean of non-missing subscales.
  score on a scale | 78.4 [33 to 98] | 78.3 [20 to 99] | 77.3 [27 to 100] | 78 [20 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Stable Vision at Week 52
Description: Stable vision was defined as vision loss of fewer than 15 letters in Best-corrected Visual Acuity (BCVA) from baseline. BCVA is measured using an eye chart and is reported as the number of letters read correctly using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. The percentage of participants with a BCVA loss of fewer than 15 letters are reported. Study eye was defined as the eye that meets the entry criteria. If both the eyes met all of the entry criteria, the eye with worse BCVA at baseline (Day 1) was selected. If BCVA values for both eyes were identical then participant had to select the non-dominant eye, or else right eye was selected as study eye.
Time Frame: Baseline to Week 52
Population: Per Protocol (PP) population included all randomized and treated participants without any protocol deviations that impacted the primary efficacy variable and with treatment compliance to represent the intended regimen adequately.
Measure: Number; unit: percentage of participants
Arm/Group | Abicipar Pegol 2 mg (2Q8) | Abicipar Pegol 2 mg (2Q12) | Ranibizumab (rQ4)
Number analyzed (Participants) | 267 | 265 | 299
percentage of participants | 94.8 | 91.3 | 96.0
Statistical Analysis 1: Comparison: Abicipar Pegol 2 mg (2Q8) vs Ranibizumab (rQ4); Test type: Non-Inferiority — For hypothesis testing, if the lower limit of the 95.1% confidence interval for the difference between an abicipar group and ranibizumab is greater than or equal to -10%, non-inferiority of abicipar group is established; Percentage Difference = -1.2, 95% CI 2-sided [-5.0 to 2.4] — The 95.1% CI for the weighted difference were calculated based on the Newcombe method using the Cochran-Mantel-Haenszel weights and baseline BCVA (≤55 vs >55 letters) as stratification factor
Statistical Analysis 2: Comparison: Abicipar Pegol 2 mg (2Q12) vs Ranibizumab (rQ4); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Percentage Difference = -4.6, 95% CI 2-sided [-9.0 to -0.5] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Mean Change From Baseline in Best-corrected Visual Acuity (BCVA) in the Study Eye at Week 52
Description: BCVA was measured using an eye chart and is reported as the number of letters read correctly using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. Mixed-effect model for repeated measures (MMRM) analysis was used. Study eye is defined as the eye that meets the entry criteria. If both the eyes met all of the entry criteria, the eye with worse BCVA at baseline (Day 1) was selected. If BCVA values for both eyes were identical then participant had to select the non-dominant eye, or else right eye was selected as study eye.
Time Frame: Baseline to Week 52
Population: PP population included all randomized and treated participants without any protocol deviations that impacted the primary efficacy variable and with treatment compliance to represent the intended regimen adequately. Number of participants analyzed was based on observed data; missing data were not imputed.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Abicipar Pegol 2 mg (2Q8) | Abicipar Pegol 2 mg (2Q12) | Ranibizumab (rQ4)
Number analyzed (Participants) | 248 | 251 | 287
letters | 8.3 (14.3) | 7.3 (13.8) | 8.3 (11.8)
Statistical Analysis 1: Comparison: Abicipar Pegol 2 mg (2Q8) vs Ranibizumab (rQ4); Test type: Non-Inferiority — For hypothesis testing, non-inferiority of abicipar is established if the lower limit of the CI is > - 5.0 letters; Least Squares Mean Difference = -0.2, 95.1% CI 2-sided [-2.4 to 2.0], Standard Error of Mean 1.1 — MMRM included treatment, region, BL BCVA, BL CRT ≤400 or >400, choroidal neovascularization lesion type, visit, visit-by-BL BCVA interaction, and treatment-by-visit interaction term as covariates using an unstructured covariance matrix
Statistical Analysis 2: Comparison: Abicipar Pegol 2 mg (2Q12) vs Ranibizumab (rQ4); Test type: Non-Inferiority — For hypothesis testing, non-inferiority of abicipar is established if the lower limit of the CI is > - 5.0 letters; Least Squares Mean Difference = -1.6, 95.1% CI 2-sided [-3.8 to 0.6], Standard Error of Mean 1.1 — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Mean Change From Baseline in Central Retinal Thickness (CRT) in the Study Eye at Week 52
Description: CRT was assessed using spectral domain optical coherence tomography (SD-OCT), a non-invasive diagnostic system that provides high-resolution imaging sections of the retina. SD-OCT is performed in the study eye after pupil dilation. A negative change from Baseline indicates improvement and a positive change from baseline indicates worsening. Study eye is defined as the eye that meets the entry criteria. If both the eyes met all of the entry criteria, the eye with worse BCVA at baseline (Day 1) was selected. If BCVA values for both eyes were identical then participant had to select the non-dominant eye, or else right eye was selected as study eye. MMRM analysis was used.
Time Frame: Baseline to Week 52
Population: Intent-to-treat (ITT) Population included all randomized participants. Number of participants analyzed was based on observed data; missing data were not imputed.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Abicipar Pegol 2 mg (2Q8) | Abicipar Pegol 2 mg (2Q12) | Ranibizumab (rQ4)
Number analyzed (Participants) | 248 | 256 | 286
microns | -146.8 (118.1) | -141.7 (127.1) | -147.1 (126.2)
Statistical Analysis 1: Comparison: Abicipar Pegol 2 mg (2Q8) vs Ranibizumab (rQ4); Test type: Superiority — Superiority of abicipar was demonstrated if the lower limit of CI for the treatment difference was greater than zero; Least Squares Mean Difference = 3.5, 95.1% CI 2-sided [-7.1 to 14.0], Standard Error of Mean 5.4 — MMRM included treatment, region, BL BCVA, BL CRT, choroidal neovascularization lesion type, visit, visit-by-baseline CRT interaction, and treatment-by-visit interaction term as covariates using an unstructured covariance matrix
Statistical Analysis 2: Comparison: Abicipar Pegol 2 mg (2Q12) vs Ranibizumab (rQ4); Test type: Superiority — Superiority of abicipar was demonstrated if the lower limit of CI for the treatment difference was greater than zero; Least Squares Mean Difference = 5.9, 95.1% CI 2-sided [-4.7 to 16.5], Standard Error of Mean 5.4 — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Percentage of Participants With BCVA Gain of More Than 15 Letters From Baseline in the Study Eye at Week 52
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly using the Early Treatment of Diabetic Retinopathy Study (ETDRS) Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. The percentage of participants with a BCVA gain of more than 15 letters are noted. Study eye is defined as the eye that meets the entry criteria. If both the eyes met all of the entry criteria, the eye with worse BCVA at baseline (Day 1) was selected. If BCVA values for both eyes were identical then participant had to select the non-dominant eye, or else right eye was selected as study eye.
Time Frame: Baseline to Week 52
Population: ITT Population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Abicipar Pegol 2 mg (2Q8) | Abicipar Pegol 2 mg (2Q12) | Ranibizumab (rQ4)
Number analyzed (Participants) | 316 | 315 | 318
percentage of participants | 28.2 | 24.4 | 26.7
Statistical Analysis 1: Comparison: Abicipar Pegol 2 mg (2Q8) vs Ranibizumab (rQ4); Test type: Superiority; Percentage Difference = 1.4, 95% CI 2-sided [-5.5 to 8.4] — The 95.1% CI for the weighted difference were calculated based on the Newcombe method using the Cochran-Mantel-Haenszel weights and baseline BCVA (≤55 vs >55 letters) as the stratification factor
Statistical Analysis 2: Comparison: Abicipar Pegol 2 mg (2Q12) vs Ranibizumab (rQ4); Test type: Superiority; Percentage Difference = -2.3, 95% CI 2-sided [-9.1 to 4.5] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Mean Change From Baseline in the National Eye Institute Visual Functioning Questionnaire-25 (NEI-VFQ-25) Composite Score at Week 52
Description: NEI-VFQ-25 consists of 25 vision-targeted questions that represent 11 vision-related quality of life subscales and one general health item. Responses of individual participants were recorded as scores that ranged between 0 (worst) to 100 (best vision related function) with higher scale indicating better vision. Overall composite score is then calculated by averaging over all 11 vision-targeted subscale scores, excluding general health score. Overall composite score was calculated based on mean of non-missing subscales. Study eye: eye that meets entry criteria. If both eyes met all of entry criteria, eye with worse BCVA at baseline (day 1) was selected. If BCVA values for both eyes were identical then participant had to select non-dominant eye, or else right eye was selected as study eye. A positive change from baseline indicates improvement. MMRM analysis was used.
Time Frame: Baseline to Week 52
Population: ITT population included all randomized participants. Number of participants analyzed was based on observed data; missing data were not imputed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Abicipar Pegol 2 mg (2Q8) | Abicipar Pegol 2 mg (2Q12) | Ranibizumab (rQ4)
Number analyzed (Participants) | 254 | 261 | 287
scores on a scale | 2.8 (0.7) | 2.4 (0.7) | 4.4 (0.7)
Statistical Analysis 1: Comparison: Abicipar Pegol 2 mg (2Q8) vs Ranibizumab (rQ4); Test type: Superiority — Superiority of abicipar was demonstrated if the lower limit of CI for the treatment difference was greater than zero; Least Squares Mean Difference = -1.6, 95.1% CI 2-sided [-3.5 to 0.3], Standard Error of Mean 1.0 — MMRM included treatment group, region, baseline BCVA in the study eye, baseline VFQ score, visit, and treatment by visit interaction as fixed covariates using an unstructured covariance matrix
Statistical Analysis 2: Comparison: Abicipar Pegol 2 mg (2Q12) vs Ranibizumab (rQ4); Test type: Superiority — Superiority of abicipar was demonstrated if the lower limit of CI for the treatment difference was greater than zero; Least Squares Mean Difference = -2.0, 95.1% CI 2-sided [-3.9 to -0.1], Standard Error of Mean 1.0 — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: From the first dose up to last dose (Up to Week 104)
Description: Safety population included all treated participants.
Arm/Group | Abicipar Pegol 2 mg (2Q8) | Abicipar Pegol 2 mg (2Q12) | Ranibizumab (rQ4)
All-Cause Mortality (participants affected / at risk) | 11/313 | 6/314 | 7/315
Serious Adverse Events (participants affected / at risk) | 94/313 | 83/314 | 78/315
Other Adverse Events (participants affected / at risk) | 168/313 | 166/314 | 166/315
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abicipar Pegol 2 mg (2Q8) (N=313) | Abicipar Pegol 2 mg (2Q12) (N=314) | Ranibizumab (rQ4) (N=315)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 3 | 5 | 5
Atrial fibrillation (Cardiac disorders) | 2 | 3 | 5
Angina pectoris (Cardiac disorders) | 1 | 2 | 3
Coronary artery disease (Cardiac disorders) | 1 | 1 | 2
Arrhythmia (Cardiac disorders) | 0 | 1 | 2
Bradycardia (Cardiac disorders) | 0 | 0 | 2
Myocardial infarction (Cardiac disorders) | 0 | 4 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Myocardial oedema (Cardiac disorders) | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 2 | 1 | 0
Aortic valve disease (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 1 | 1
Meniere's disease (Ear and labyrinth disorders) | 0 | 1 | 0
Retinal haemorrhage (Eye disorders) | 2 | 0 | 5
Retinal detachment (Eye disorders) | 3 | 0 | 2
Cataract (Eye disorders) | 2 | 3 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 2 | 1
Retinal fibrosis (Eye disorders) | 0 | 0 | 1
Retinal pigment epithelial tear (Eye disorders) | 0 | 0 | 1
Uveitis (Eye disorders) | 7 | 4 | 0
Retinal vasculitis (Eye disorders) | 4 | 4 | 0
Visual acuity reduced (Eye disorders) | 1 | 3 | 0
Vitritis (Eye disorders) | 4 | 1 | 0
Iridocyclitis (Eye disorders) | 2 | 1 | 0
Retinal artery occlusion (Eye disorders) | 1 | 1 | 0
Age-related macular degeneration (Eye disorders) | 0 | 1 | 0
Autoimmune uveitis (Eye disorders) | 0 | 1 | 0
Choroidal neovascularisation (Eye disorders) | 0 | 1 | 0
Neovascular age-related macular degeneration (Eye disorders) | 0 | 1 | 0
Retinal vein occlusion (Eye disorders) | 0 | 1 | 0
Anterior chamber inflammation (Eye disorders) | 1 | 0 | 0
Keratitis (Eye disorders) | 1 | 0 | 0
Macular hole (Eye disorders) | 1 | 0 | 0
Serous retinal detachment (Eye disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 3 | 8
Diverticulitis (Infections and infestations) | 0 | 1 | 2
Endophthalmitis (Infections and infestations) | 5 | 4 | 1
Sepsis (Infections and infestations) | 2 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 1
Arteritis infective (Infections and infestations) | 0 | 0 | 1
Enterocolitis viral (Infections and infestations) | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1
Infective aortitis (Infections and infestations) | 0 | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Pneumonia escherichia (Infections and infestations) | 0 | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 3 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Infectious colitis (Infections and infestations) | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 3 | 3
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 1
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 1
Intraocular pressure increased (Investigations) | 1 | 2 | 0
Heart rate decreased (Investigations) | 0 | 1 | 0
Monoclonal immunoglobulin present (Investigations) | 0 | 1 | 0
Blood glucose abnormal (Investigations) | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0
Pulmonary function test decreased (Investigations) | 1 | 0 | 0
Urine electrolytes decreased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Bone loss (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Foot fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 6
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Retroperitoneal neoplasm metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 3
Cerebrovascular accident (Nervous system disorders) | 0 | 3 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1
Brain stem stroke (Nervous system disorders) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Piriformis syndrome (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Optic neuritis (Nervous system disorders) | 0 | 1 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 1 | 0
Vertebral artery occlusion (Nervous system disorders) | 0 | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Speech disorder (Nervous system disorders) | 1 | 0 | 0
Vascular dementia (Nervous system disorders) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 2
Aortic stenosis (Vascular disorders) | 0 | 1 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 2 | 0
Blood pressure inadequately controlled (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0
Peripheral artery aneurysm (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abicipar Pegol 2 mg (2Q8) (N=313) | Abicipar Pegol 2 mg (2Q12) (N=314) | Ranibizumab (rQ4) (N=315)
Eye pain (Eye disorders) | 37 | 35 | 36
Conjunctival haemorrhage (Eye disorders) | 24 | 29 | 29
Conjunctival hyperaemia (Eye disorders) | 17 | 15 | 23
Neovascular age-related macular degeneration (Eye disorders) | 18 | 25 | 21
Vitreous floaters (Eye disorders) | 27 | 30 | 17
Vitreous detachment (Eye disorders) | 16 | 17 | 11
Visual acuity reduced (Eye disorders) | 17 | 15 | 6
Nasopharyngitis (Infections and infestations) | 33 | 35 | 40
Influenza (Infections and infestations) | 19 | 15 | 22
Urinary tract infection (Infections and infestations) | 22 | 21 | 12
Fall (Injury, poisoning and procedural complications) | 13 | 14 | 22
Intraocular pressure increased (Investigations) | 29 | 29 | 20
Headache (Nervous system disorders) | 11 | 18 | 17
Hypertension (Vascular disorders) | 18 | 22 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT02462486/SAP_000.pdf
  • Study Protocol (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/86/NCT02462486/Prot_001.pdf